CLINICAL TRIAL: NCT02699892
Title: Post Marketing Non Interventional Clinical Research of Administration of Rituximab in Rheumatoid Arthritis
Brief Title: Study to Examine Efficacy and Safety of Rituximab in Participants With Rheumatoid Arthritis
Acronym: RITAM
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21619
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid arthritis participants: Participants who were on rituximab for rheumatoid arthritis and who will continue receiving rituximab treatment (at the discretion of treating physician) according to previous approved indication will be observed for a period of 72 weeks.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered at the discretion of treating physician according to approved label. Protocol does not specify/enforce the criteria for initiation of treatment with rituximab and procedure of the infusion of rituximab.
  Other Names: MabThera

SUMMARY:
This Phase IV post-marketing, non-interventional, open label, non-comparative and prospective study will examine the efficacy and safety of rituximab in participants who had previously received rituximab in terms of everyday medical practice. Efficacy and safety of rituximab will be determined 24 weeks after receiving the first infusion, 24 weeks after the second infusion repeated courses of treatment (if the participants receive another course of rituximab) and 24 weeks after the third infusion repeated courses of treatment (if the participants receive third course of rituximab). Protocol does not specify the criteria for initiation of treatment with rituximab and procedure of the infusion of rituximab. Rituximab will be administered at the discretion of treating physician according to approved label.

ELIGIBILITY:
Inclusion Criteria:

-Participants receiving rituximab no longer than 4 weeks before the start of monitoring

Exclusion Criteria:

-Not Applicable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving rituximab no longer than 4 weeks for the treatment of rheumatoid arthritis before the start of study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2007-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Serbia (4):
  - Belgrade
  - Niška Banja
  - Nova Sad
  - Novi Sad

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no documentation for the reason for discontinuation; hence, in Participant Flow module, for all participants who did not complete the study, the reason is reported as Unspecified.
Groups:
- Rheumatoid Arthritis Participants: Participants who were on rituximab for rheumatoid arthritis and who continued receiving rituximab treatment (at the discretion of treating physician) according to approved label were observed for a period of 72 weeks.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Participants
Started | 130
Completed | 94
Not Completed | 36
Not completed — Other | 36

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants, who received at least one dose of the drug under observation and had a subsequent post baseline assessment.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.28 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Reduction From Baseline in Disease Activity Score Based on 28 Joints Count (DAS28) of More Than 1.2 Units After 24 Weeks of First Rituximab Infusion
Description: DAS28 score is a measure of participant's disease activity calculated using tender joint count [28 joints] (TJC28), swollen joint count [28 joints] (SJC28), participant's global assessment of disease activity (PGH) [visual analog scale (VAS): 0=no disease activity to 100=maximum disease activity] and erythrocyte sedimentation rate (ESR). DAS28 was calculated according to following formula: [0.56 multiplied by (*) square root (√) of TJC] plus (+) [0.28*√SJC]+[0.70*the natural logarithm (ln) ESR]+[0.014*PGH]. Total possible score of 0 to approximately 10, where higher scores represented higher disease activity. Scores below 2.6 indicated clinical remission, score of less than or equals to (</=) 3.2 indicated low disease activity, score of greater than (>) 3.2 to </=5.1 indicated moderate disease activity, scores above 5.1 indicated high or severe disease.
Time Frame: Baseline, 24 weeks after first rituximab infusion (Week 24)
Population: ITT population. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 112
Percentage of participants | 61.60

2. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Good Response
Description: Clinical response was assessed according to EULAR categorical DAS28 response criteria, which defined clinically meaningful improvement at Weeks 24, 48, and 72. EULAR response was based on change from baseline (CFB) in DAS28 score and on actual DAS28 score, at Weeks 24, 48, and 72. DAS28 score: participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. DAS28 was calculated by following formula: (0.56*√TJC)+(0.28*√SJC)+(0.70*ln ESR)+(0.014*PGH). Total possible score = 0-10, higher scores represented higher disease activity. EULAR Good response: DAS28</=3.2; reduction of DAS28 >1.2.
Time Frame: Baseline, Weeks 24, 48 and 72
Population: ITT Population. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome and "n" signified those participants who were evaluable for a specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 112
Percentage of participants
  Week 24 (n=112) | 21.43
  Week 48 (n=81) | 16.05
  Week 72 (n=59) | 18.64

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (up to 72 weeks )
Description: Safety population included all participants who received at least one dose of drug under observation and had a subsequent safety assessment.
Arm/Group | Rheumatoid Arthritis Participants
Serious Adverse Events (participants affected / at risk) | 11/130
Other Adverse Events (participants affected / at risk) | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=130)
Drug hypersensitivity (Immune system disorders) | 4
Urticaria (Immune system disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Streptococcal sepsis (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Gastritis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Pyelonephritis acute (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.